CLINICAL TRIAL: NCT00514267
Title: A Phase I/II Multicenter, Open-Label Study of YM155 Plus Docetaxel in Subjects With Advanced Hormone Refractory Prostate Cancer and Other Solid Tumors
Brief Title: An Open-Label Study of YM155 + Docetaxel in Subjects With Advanced Hormone Refractory Prostate Cancer and Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-025
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Prostate Cancer; Tumors
Keywords: Prostate Cancer; HRPC; Hormone Refractory Prostate Cancer; YM155; Treatment Outcome; Solid Tumors
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — sepantronium; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. HRPC (Experimental)
  Interventions: Drug: YM 155; Drug: Docetaxel; Drug: Prednisone
- 2. Solid Tumors (Experimental)
  Interventions: Drug: YM 155; Drug: Docetaxel

INTERVENTIONS:
Drug: YM 155 — IV
Drug: Docetaxel — IV
Drug: Prednisone — Oral
  Arms: 1. HRPC

SUMMARY:
To determine the feasibility and safety of administering YM155 in combination with docetaxel

DETAILED DESCRIPTION:
This clinical trial is designed to include two parts:

Part 1: Assessment of feasibility and safety of administering YM155 in combination with docetaxel and prednisone in subjects with hormone refractory prostate cancer (HRPC) [ ENROLLMENT COMPLETED ]

Part 2: Assessment of feasibility and safety of administering YM155 in combination with docetaxel in subjects with solid tumors (except HRPC).

This registration has been updated to reflect the design requirements of PART 2.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Male subjects with histologically or cytologically confirmed adenocarcinoma of the prostate with clinical or radiological evidence of metastatic disease.

Part 2:

* Subjects with histologically and cytologically confirmed solid tumors with measurable disease (except HRPC).

Exclusion Criteria:

* Radiation therapy within 4 weeks of the start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (Part 1: Subjects with HRPC) | 2 cycles
Occurrence of dose limiting toxicities (Part 2: Subjects with other solid tumors) | 1 cycle

SECONDARY OUTCOMES:
Assessment of safety and efficacy | 10 cycles
Assessment of pharmacokinetics | Part 1 only

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- San Antonio, Texas, United States